CLINICAL TRIAL: NCT03992768
Title: Clinical Validation for Feature Detection Precision by WSI Using Hamamatsu NanoZoomer S360MD Digital Slide Scanner System
Brief Title: Feature Detection Study for Validation of Hamamatsu NanoZoomer S360MD Digital Slide Scanner System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamamatsu Photonics K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCT-P002
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Pathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NanoZoomer Whole Slide Imaging (Experimental): Whole slide imaging using the Hamamatsu NanoZoomer S360MD Digital Slide Scanner System
  Interventions: Device: Hamamatsu NanoZoomer S360MD Digital Slide Scanner System

INTERVENTIONS:
Device: Hamamatsu NanoZoomer S360MD Digital Slide Scanner System — Detection of pathology features using whole slide imaging

SUMMARY:
The objective of this study is to evaluate the repeatability and reproducibility of detection of histological features using whole slide imaging

DETAILED DESCRIPTION:
The study will be conducted under the following 3 sub-studies:

1. Scans within Scanner (Intra-scanner precision substudy),
2. Scanners within a site (Inter-scanner precision substudy),
3. Scanners between sites (Inter-site precision substudy)

ELIGIBILITY:
Inclusion Criteria:

Glass slides are screened for the known features and will be considered eligible for the study only if all of the following criteria apply:

* Slides are selected from cases in a consecutive manner starting with cases at least 1 year old since accessioning
* Slide is a glass cover-slipped surgical pathology slide of human tissue
* Slide is stained with hematoxylin and eosin (H&E) or other stains
* Slide has the designated primary feature in the FOV, which is readily observable in its natural environment although the slide may also have one or more secondary features from the same magnification group in the FOV.
* Slide is available in the archives for use, or purchased commercially, is not damaged, has tissue on the slide which is still in good condition, has a stain that is not faded and otherwise passes all quality checks

Exclusion Criteria:

Slides are to be excluded from the study if any of the following criteria apply:

* Slide is unable to be scanned, contains damaged tissue or has indelible markings
* Slide comes from an active (less than 1 year old) case
* Slide is from a patient who already has a slide enrolled in the study, only 1 slide per patient to be enrolled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Parwani, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Washington University, St Louis, Missouri
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Features
Period: Overall Study
Arm/Group | NanoZoomer Whole Slide Imaging
Started | 540; 540 Features
Completed | 540; 540 Features
Not Completed | 0; 0 Features

BASELINE CHARACTERISTICS:
Arm/Group | NanoZoomer Whole Slide Imaging
Number analyzed (Participants) | 540
Age, Categorical [Count of Participants; unit: Participants] — These data were not collected in this study. Population: Due to the fact that no subject-specific information was required for this study, no demographic information was collected.
Sex: Female, Male [Count of Participants; unit: Participants] — These data were not collected in this study. Population: Due to the fact that no subject-specific information was required for this study, no demographic information was collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 540

OUTCOME MEASURES:

1. Primary Outcome: Overall Percentage Agreement of Repeatability and Reproducibility Within Scanner, Between Scanners, and Sites.
Description: Repeatability and reproducibility of WSI were evaluated using the Average Positive Agreement Rate. Using a comparison of two reads with four possible outcomes (a=both reads detect the feature; b=read 1 fails to detect the feature; c=read 2 fails to detect the feature; d=both reads fail to detect the feature), APA = 2a/(2a+b+c). APA was used to assess outcomes in the following substudies:
  1. Scans within scanner (Intra-scanner Precision): Scans are repeated within the scanner at the site.
  2. Scanners within site (Inter-scanner Precision): Scans are repeated among the scanners at the site
  3. Scans between Sites (Inter-site Precision): Scans are repeated within the scanner at the different sites.
Time Frame: 1 day
Population: Intra-scanner Precision: 3 separate scans on 1 scanner of 378 features read by 3 reading pathologists in 3 sessions each Inter-scanner Precision: 1 scan each of 378 features on 3 scanners read by 3 reading pathologists in 3 sessions each Inter-site Precision: 378 FOVs scanned on 1 scanner read by 3 reading pathologists at 3 sites in 1 session each
Measure: Number (95% Confidence Interval); unit: Average Positive Agreement Rate
Units Other Than Participants: Reads
Groups:
- NanoZoomer Whole Slide Imaging - Intra-scanner Precision; NanoZoomer Whole Slide Imaging - Inter-scanner Precision; NanoZoomer Whole Slide Imaging - Inter-site Precision: Hamamatsu NanoZoomer S360MD Digital Slide Scanner System: Detection of pathology features using whole slide imaging
Arm/Group | NanoZoomer Whole Slide Imaging - Intra-scanner Precision | NanoZoomer Whole Slide Imaging - Inter-scanner Precision | NanoZoomer Whole Slide Imaging - Inter-site Precision
Number analyzed (Participants) | 540 | 540 | 540
Number analyzed (Reads) | 3402 | 3402 | 1134
Average Positive Agreement Rate | 94.5 [93.7 to 95.3] | 92.4 [90.7 to 93.9] | 93.4 [91.9 to 94.9]

ADVERSE EVENTS:
Time Frame: Because there was no patient involvement in the study and no impact on patient diagnoses, there were no safety endpoints for the study
Description: Because there was no patient involvement in the study and no impact on patient diagnoses, there were no safety endpoints for the study. Hence, there was no monitoring or assessment for adverse events
Arm/Group | NanoZoomer Whole Slide Imaging
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT03992768/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03992768/SAP_001.pdf